CLINICAL TRIAL: NCT05778838
Title: Clinical Study Evaluating the Efficacy and Safety of Adjunctive Use of Midodrine in Septic Shock Patients
Brief Title: Midodrine Effect on the Mortality Rates in Septic Shock Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noha Mansour (Other)
Responsible Party: Sponsor-Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-211
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Will receive IV vasopressor infusion only
  Interventions: Drug: Midodrine Oral Tablet
- Midodrine (Active Comparator): Will receive oral midodrine 10 mg/ 8 hours in addition to IV vasopressor infusion till the end of treatment (subject remaining vasopressor-free for 24 consecutive hours).
  Interventions: Drug: Midodrine Oral Tablet

INTERVENTIONS:
Drug: Midodrine Oral Tablet — Patients will receive standard treatment in accordance to surviving sepsis campaign guidelines plus oral midodrine 10 mg/ 8 hours till the end of treatment (subject remaining vasopressor-free for 24 consecutive hours) or death.

SUMMARY:
Assessing the safety and efficacy of the adjunctive use of midodrine as a vasopressor in septic shock patients by measuring the difference in the mortality rates between control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or older diagnosed with septic shock.
* Hypotensive and require IV vasopressor for more than 24 hours.

Exclusion Criteria:

* Hypovolemic shock.
* Severe organic heart disease (ejection fraction <30 percent).
* Bradycardia (HR<50 b/m).
* Chronic kidney disease (serum creatinine >2mg/dl).
* Thyrotoxicosis.
* Pheochromocytoma.
* Known allergy to midodrine.
* Unable to administer an oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Mortality rates | Time Frame: Starting from date of randomization till shock reversal or date of death from any cause, whichever came first,assessed up to 30 days
  The primary outcome is measuring the difference in ICU mortality rates between control and intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No